CLINICAL TRIAL: NCT02432651
Title: Prevention of Oxidative DNA Damage by Xanthohumol
Brief Title: Xanthohumol and Prevention of DNA Damage
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Oregon State University (Other)
Responsible Party: Principal Investigator, Jan Frederik Stevens, Professor of Medicinal Chemistry, Department of Pharmaceutical Sciences, College of Pharmacy, Oregon State University
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LPI-6119
Record Dates: First submitted 2015-03-09; First posted 2015-05-04 (Estimated); Last update posted 2018-11-06 (Actual); Status verified 2018-11

CONDITIONS: Oxidative Stress
Keywords: oxidative stress; hops; xanthohumol; DNA damage; cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 6 mg xanthohumol per day vs. placebo (Other): All participants take 6 mg xanthohumol daily and placebo in a crossover design with a washout period.
  Interventions: Drug: 6 mg xanthohumol per day; Drug: Placebo
- 12 mg xanthohumol per day vs. placebo (Other): All participants take 12 mg xanthohumol daily and placebo in a crossover design with a washout period.
  Interventions: Drug: 12 mg xanthohumol per day; Drug: Placebo
- 24 mg xanthohumol per day vs. placebo (Other): All participants take 24 mg xanthohumol daily and placebo in a crossover design with a washout period.
  Interventions: Drug: 24 mg xanthohumol per day; Drug: Placebo

INTERVENTIONS:
Drug: 6 mg xanthohumol per day — Participants will consume non-alcoholic beverage with 2 mg xanthohumol at breakfast, lunch and dinner for 3 weeks.
  Arms: 6 mg xanthohumol per day vs. placebo
Drug: 12 mg xanthohumol per day — Participants will consume a non-alcoholic beverage with 2 mg xanthohumol at breakfast and lunch and 8 mg at dinner for 3 weeks.
  Arms: 12 mg xanthohumol per day vs. placebo
Drug: 24 mg xanthohumol per day — Participants will consume a non-alcoholic beverage with 8 mg xanthohumol at breakfast, lunch and dinner for 3 weeks.
  Arms: 24 mg xanthohumol per day vs. placebo
Drug: Placebo — Participants will consume a placebo non-alcoholic beverage (0 mg xanthohumol) at breakfast, lunch and dinner for 3 weeks.

SUMMARY:
The purpose of this research study is to learn if and in what amount a compound from hops, called xanthohumol (ZAN-tho-HUE-mol), prevents damage to DNA and oxidative stress. The human body is constantly exposed to oxidative stress from environmental compounds (e.g. air pollution) which may cause damage to DNA. The human body can repair some DNA damage, but too much DNA damage is harmful and may lead to cancer. Research done at OSU and around the world has shown that xanthohumol can stop or slow processes that lead to cancer.

DETAILED DESCRIPTION:
The purpose of this research study is to learn if and in what amount a compound from hops, called xanthohumol (ZAN-tho-HUE-mol), prevents damage to DNA and oxidative stress. The human body is constantly exposed to oxidative stress from environmental compounds (e.g. air pollution) which may cause damage to DNA. The human body can repair some DNA damage, but too much DNA damage is harmful and may lead to cancer. Research done at OSU and around the world has shown that xanthohumol can stop or slow processes that lead to cancer.

Participants will consume a non-alcoholic beverage containing xanthohumol with breakfast, lunch and dinner for 3 weeks. Then they will go through a washout period of 3 weeks. And then they will consume the same beverage without the xanthohumol compound (placebo) for another 3 weeks. Participants will be randomly assigned into groups and will vary whether they will consume the xanthohumol product during the first or second 3-week period. Xanthohumol doses will be 0, 6, 12 or 24 mg/day.

The study includes donation of blood and urine samples and one-month food frequency questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Non-smokers or no other tobacco use in the past 3 months.
* Willing to stop taking regular supplements including anti-oxidants for 2 weeks prior to study entry through conclusion of study.
* Willing to stop consumption of high levels of flavonoids and xanthohumol in the normal diet (onions, teas including green/black tea and microbrew beers) for 2 weeks prior to study entry through conclusion of study.
* Must be able to give written informed consent.
* Blood screen tests (Comprehensive metabolic profile [CMP] and lipid profile) within normal limits.

Exclusion Criteria:

* Body Mass Index (BMI) less than 18.5 (underweight) or greater than 30 (obese)
* Have a significant acute or chronic coexisting illness such as cardiovascular disease, chronic kidney or liver disease, gastrointestinal disorder, endocrinological disorder, immunological disorder, metabolic disease, cancer, history of chemotherapy, celiac disease or gluten/wheat intolerance*, diabetes, thyroid problems, or any condition which contraindicates, in the investigators judgement, entry into the study.
* Currently taking prescription drugs except oral contraceptives.
* Consumption of more than the recommended alcohol guidelines i.e. >2 drinks/day.
* Consumption of high levels of flavonoids and xanthohumol in the normal diet (onions, teas including green/black tea and microbrew beers).
* Pregnancy (as confirmed by urine pregnancy test), breastfeeding, or planning to become pregnant before completing the study.
* Undergoing UV therapy (e.g. treatment for skin conditions such as psoriasis), using UV tanning beds, or unprotected sun exposure greater than 1 hour per day.
* Engaging in vigorous exercise more than 6 hours per week.
* Participation in another dietary study in the past 3 months.
* Had surgery in the last 3 months.
* Post-menopausal status

(*Note: Beverage is formulated with a barley extract. Barley contains gluten.)

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 64 (Actual)
Dates: Start 2015-03; Primary Completion 2016-06 (Actual); Study Completion 2017-06 (Actual)

PRIMARY OUTCOMES:
Comparison of the change in markers of DNA damage and oxidative stress during XN treatment vs. the change during placebo | Prior to first dose on day 1 to day 63.
  Plasma and urine levels of 8-oxo-dG will be measured at the beginning and end of each 3-week cycle. DNA strand breaks in blood cells and plasma levels of reduced and oxidized glutathione will be measured at the beginning and end of each 3-week cycle. Between the two cycles, there will be a 3-week washout. One cycle is XN treatment, and one cycle is the placebo.

SECONDARY OUTCOMES:
Comparison of the change in metabolic profile during XN treatment vs. the change during placebo | Prior to first dose on day 1 to day 63.
  Metabolome measurements in plasma at beginning and end of first 3-week cycle with 3-week. Between the two cycles, there will be a 3-week washout period between cycles. One cycle is XN treatment, and one cycle is the placebo.

CONTACTS AND LOCATIONS:
Overall Officials: Jan Frederik Stevens, PhD, Principal Investigator — Oregon State University
Locations (1):
- Oregon State University, Corvallis, Oregon, United States

IPD SHARING:
Plan to Share IPD: No